CLINICAL TRIAL: NCT03191981
Title: A Phase I/II Trial Investigating the Combination of Pembrolizumab (Keytruda) With Cyclophosphamide and Lenalidomide for Patients With Relapsed Multiple Myeloma
Brief Title: Pembrolizumab Cyclophosphamide and Lenalidomide for Patients With Relapsed Multiple Myeloma
Acronym: MUKfourteen
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawal of pharma support prior to opening to recruitment
Sponsor: University of Leeds (Other)
Collaborators: Myeloma UK (Other); Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM16/87650
Record Dates: First submitted 2017-05-24; First posted 2017-06-19 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Myeloma Multiple
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; Lenalidomide; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase I/II trial with an initial dose finding phase for cyclophosphamide and lenalidomide combined with fixed dose pembrolizumab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Cyclophosphamide and lenalidomide combined with fixed dose pembrolizumab
  Interventions: Drug: Cyclophosphamide; Drug: Lenalidomide; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Cyclophosphamide — Treatment for all patients will be with cyclophosphamide, lenalidomide and pembrolizumab at fixed doses.
Drug: Lenalidomide — Treatment for all patients will be with cyclophosphamide, lenalidomide and pembrolizumab at fixed doses.
  Other Names: Revlimid
Drug: Pembrolizumab — Treatment for all patients will be with cyclophosphamide, lenalidomide and pembrolizumab at fixed doses.
  Other Names: Keytruda

SUMMARY:
This is a multi-centre phase I/II trial with an initial dose finding phase for cyclophosphamide and lenalidomide combined with fixed dose pembrolizumab for patients with relapsed or relapsed / refractory multiple myeloma (MM) that have had at least 1 prior line of therapy

DETAILED DESCRIPTION:
This is a multi-centre phase I/II trial with an initial dose finding phase for cyclophosphamide and lenalidomide combined with fixed dose pembrolizumab for patients with relapsed or relapsed / refractory MM that have had at least one prior line of therapy.

As this combination has not been given before, participants will be registered initially into a dose finding phase where dose limiting toxicities (DLTs) will be monitored during the first cycle in order to confirm the recommended dose schedule (RD) of cyclophosphamide with lenalidomide and fixed dose pembrolizumab. A modified toxicity probability interval (mTPI) approach has been taken for dose finding, to determine a safe dose schedule defined as the probability of dose limiting toxicity below an acceptable rate of 34%.

Once a RD is identified an expansion phase is planned to estimate the activity profile of the Key-CR combination at the RD. The trial will start at the highest dose schedule . Cohorts of 3 evaluable participants will sequentially be recruited to the trial until the RD has been identified or the trial stopped due to excessive toxicity at dose schedule -1. The dose schedule to be given to a subsequent cohort will be evaluated after all participants have been followed up for one cycle or experienced a DLT. The Safety Review Committee (SRC) will be presented with a complete safety report in addition to a set of predetermined dosing decisions, such that all relevant information available may be considered before deciding upon the next dose schedule to be allocated.

The mTPI is an adaptive Bayesian design specifying that the parameter for the probability that a patient experiences a DLT during the first cycle follows a separate distribution for each dose level. Each DLT probability is believed to be equally likely to take any value between 0 and 1 before any data is collected this represents a non-informative or flat prior. The posterior distribution from which escalation decisions are made is constructed by updating the prior distribution with observed data and represents our updated beliefs about the parameter after having seen the data. The decision to remain at the current dose schedule (S), escalate (E), or de-escalate (D) from the posterior distribution is determined by probability theory and two clinical criteria; the minimum DLT rate that if true would warrant escalation and the maximum DLT rate that if true would warrant dose de-escalation. The clinical interval is specified to be (0.2, 0.34) in this setting. Below 0.2 would represent under-dosing and warrant escalation, above 0.34, over-dosing and de-escalation and in the interval proper dosing and the decision to remain at the current dose level.

Participants will be registered to a dose schedule in cohorts of 3 evaluable participants and a decision regarding expansion or dose (de)escalation will be made once all patients have been followed up for the full DLT observation period (see below).

A minimum of 6 participants must be evaluated at a dose schedule for the dose schedule to be considered the RD. If dose schedule -1 or 0 meet the RD criterion but the dose schedule above has not been excluded, a further cohort of participants may be treated at the dose schedule above at discretion of the SRC. If dose schedule -1 is found to be unsafe the trial will terminate early without opening the expansion phase. The SRC may consider increasing the size of cohorts after 12 evaluable participants have been treated at a dose schedule without identifying the RD. Once the RD has been identified the trial will move into the expansion phase.

It is essential that the data for each participant is returned in a timely manner to allow the participants to be monitored for safety and dose limiting toxicities that could affect the safety of other participants. Data must be returned on time to allow a timely review of the trial by the Safety Review Committee to prevent a hold up in progressing the trial to the next phase or dose level, or to allow it to be stopped quickly in the event of an unforeseen issue occurring.

Dose Schedules - 28 days schedule Dose schedule 1 (starting dose) Pembrolizumab 200mg every 3 weeks, cyclophosphamide 500mg days 1&8, lenalidomide 25mg days 1-21 Dose schedule 0 Pembrolizumab 200mg every 3 weeks, cyclophosphamide 500mg day 1, lenalidomide 25mg days 1-21 Dose schedule -1 Pembrolizumab 200mg every 3 weeks, cyclophosphamide 500mg day 1, lenalidomide 15mg days 1-21

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial and willing to follow the trial protocol.
* Be 18 years of age or greater on day of signing informed consent.
* Measurable disease with at least one of the following:

  * Paraprotein greater than or equal to 5g/L
  * Serum free light chains greater than or equal to 100mg/L with abnormal radio for light chain only
  * myeloma
  * Bence Jones protein greater than or equal to 200mg/24hr
* Have relapsed MM following 1 or more prior lines of therapy.
* Have achieved a partial response (PR or better based on investigator's determination of response by the International Myeloma Working Group (IMWG) criteria) to at least one prior regimen
* Have a performance status of 0-1 on the ECOG Performance Scale.
* Demonstrate adequate organ function as defined below, all screening laboratory tests are to be performed within 10 days prior to registration:

Haematological

* Absolute neutrophil count greater than or equal to 1.0 x109 /L. Growth factor support is not permitted within 7 days prior to assessment
* Platelet count greater than or equal to 75 x 109/L. Platelet support is not permitted within 7 days prior to assessment.
* Haemoglobin greater than or equal to 90 g/L. Blood support is not permitted within 7 days prior to assessment.

Renal

* Serum creatinine or, measured or calculated creatinine clearance less than or equal to 1.5 x local ULN OR Creatinine Clearance greater than or equal to 60 mL/min for participant with creatinine levels greater than 1.5 x local ULN Hepatic
* Serum bilirubin less than or equal to 1.5 x local ULN OR direct bilirubin less than or equal to local ULN for participants with total bilirubin levels greater than 1.5 x local ULN
* Aspartate transaminase (AST) or Alanine transaminase (ALT) less than or equal to 2.5 x local ULN
* Albumin greater than or equal to 2.5 mg/dL (25 g/L) Coagulation
* International Normalized Ratio (INR) or Prothrombin Time (PT) less than or equal to1.5 x local ULN, unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

  • The standard Celgene Revlimid REMS program must be followed for all participants taking part in the trial and followed accordingly. In addition the following must also be followed:
* Female participant of childbearing potential should have a negative urine or serum pregnancy test. Female participants of childbearing potential must be willing to use adequate methods of contraception, from 4 weeks prior to the start of treatment, until 120 days after the last dose of trial medication, and for all interruptions in dosing during the trial.
* Male participants of childbearing potential must agree to use adequate methods of contraception from 4 weeks prior to the start of treatment, until 120 days after the last dose of trial medication, and for all interruptions in dosing during the trial.

  * All participants must agree to refrain from donation blood while on trial drug, including during dose interruptions and for 120 days after discontinuation from this trial

Exclusion Criteria

* Those with non-measurable disease, solitary bone or solitary extramedullary plasmacytoma, plasma cell leukaemia, POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Is currently participating and receiving trial therapy, or has participated in a trial of an investigational agent and received trial therapy or used an investigational device within 28 days prior to the first dose of trial treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment. Steroids for myeloma disease control must be stopped 14 days prior to the first dose of trial treatment.
* If previously treated with a lenalidomide-containing regimen, the participant is excluded if:

  * Discontinued due to any adverse event related to prior lenalidomide (history of thromboembolism due to lenalidomide is allowed if participant is anticoagulated)
  * If the participant was intolerant to lenalidomide.
  * If the participant was refractory to any dose of lenalidomide. Refractory to lenalidomide is defined either:

Participant had disease progression within 60 days after the last dose of lenalidomide; or Whose disease is non-responsive whilst on lenalidomide. Non-responsive disease is defined as either not achieving at least an minimal response (MR) or progressive disease (PD) whilst on lenalidomide.

* Any of the following prior treatments:
* Has had a prior allogenic stem cell transplant. Previous autologous stem cell transplantation is permitted greater than or equal to 3 months prior to the first dose of trial treatment.
* Previous therapy with pembrolizumab or has received prior therapy with an anti-PD-1, L1 or L2 inhibitor.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to the first dose of trial treatment or who has not recovered (i.e., less than or equal to Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.

  o Has had prior chemotherapy, targeted small molecule therapy, therapeutic radiation therapy within 2 weeks prior to the first dose of trial treatment or who has not recovered (i.e., less than or equal to Grade 1 or at baseline) from adverse events due to a previously administered agent. Participants with less than ore equal to Grade 2 neuropathy are an exception to this criterion and may participant in the trial.
* Treatment with plasmapheresis within 4 weeks prior to the first dose of trial treatment.
* Palliative radiotherapy for pain control and bisphosphonates are permitted
* A known hypersensitivity or intolerance to cyclophosphamide or lenalidomide or any of its excipients.
* If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Unable to tolerate thromboembolic prophylaxis including, as clinically indicated, aspirin, warfarin or low-molecular weight heparin.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) myeloma and/or carcinomatous meningitis. Participants with previously treated CNS myeloma may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging CNS disease, and are not using steroids for at least 14 days prior to the first dose of trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Significant cardiac disease as determined by the investigator including:

  * Known or suspected cardiac amyloidosis
  * Congestive heart failure of Class III or IV of the New York Heart Association (NYHA) classification;
  * Uncontrolled angina, hypertension or arrhythmia
  * Myocardial infarction in past 6 months
  * Any uncontrolled or severe cardiovascular disease
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has an active infection requiring systemic therapy.
* Has a known history of active TB (Bacillus Tuberculosis)
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 28 days prior to the first dose of trial treatment.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.

* Is pregnant or breastfeeding, or expecting to conceive or father children within the duration of their involvement in the trial, starting with the 4 weeks prior to starting trial treatment, during trial treatment including during any treatment interruptions until 120 days after the last dose of trial treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) in dose finding phase | End of cycle 1 of treatment, 4 weeks
  Number of participants experiencing DLTs within the first cycle of treatment
Response rate | From registration until disease progression, 2 years
  Overall response rate to treatment

SECONDARY OUTCOMES:
Safety of trial treatment | From registration until the end of the trial, 2 years
  The proportion of patients experiencing at least one serious adverse event (SAE) summarising causality and seriousness.
Progression free survival (PFS) | From registration to 6 & 12 months
  The proportion of patients being progression free
Maximum response | From the start of treatment until the end of treatment, 2 years
  Maximum response achieved in response to treatment
Duration of response | From start of treatment until disease progression, 2 years
  Time for which a response to treatment was seen
Compliance to therapy | From start of treatment until the end of treatment, 2 years
  Number of patients requiring delays and/or dose reductions, treatment withdrawals.
Toxicity of trial treatment | From start of treatment until the end of treatment, 2 years
  Adverse events seen during treatment, indicating toxicity of treatment

OTHER OUTCOMES:
Overall survival | 12 months post registration
  Time to death for patients treated at the recommended dose
Time to next treatment | From end of treatment until starting the next treatment, 2 1/2 years
  Time from completing the trial treatment until next treatment is initiated for patients treated at the recommended dose

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Popat, Principal Investigator — University College, London
Locations (4):
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - University College Hospital, London
  - Guys and St Thomas NHS Foundation Trust, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
To be disseminated by trial publication and a final report